CLINICAL TRIAL: NCT06223581
Title: Evaluation of Cardiac Burden in Patients With Sever Bronchial Asthma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Hany Anwer Ahmed, Principal investigator, Assiut University
Other Study IDs: Cardiac burden in sever asthma
Record Dates: First submitted 2023-11-22; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Evaluation of Cardiac Burden in Patients With Sever Bronchial Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ECHO in sever asthma patient — Evaluation of cardiac burden in patients with sever bronchial asthma

SUMMARY:
Evaluation of cardiac burden in patients with sever bronchial asthma

DETAILED DESCRIPTION:
Bronchial asthma is chronic bronchial inflammation of variable intensity accompanied by recurrent reversible airflow obstruction and symptoms such as coughing, wheezing, shortness of breath, and chest tightness ,with a worldwide increase over the last several decades (1).

1. Sever asthma :means that asthma is uncontrolled despite adherence with maximal optimized therapy and treatment contributory factors or that worsens when high dose treatment is reduced.
2. Globally. over 260 million people had poorly controlled asthma highest rate on Australia.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted to be involved in the study.
* Patients >18 years old .

Exclusion Criteria:

* severe bronchial asthma patients who have other comorbidities as (chronic chest disease as COPD,ILD, bronchiectasis , , diabetic ,hypertensive ,mechanical ventilated patients, tracheostomized patients, ……)
* patients <18 years old . patients refuse to be involved in the study .

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Bronchial asthma is chronic bronchial inflammation of variable intensity accompanied by recurrent reversible airflow obstruction and symptoms such as coughing, wheezing, shortness of breath, and chest tightness ,with a worldwide increase over the last several decades .
  1. Sever asthma :means that asthma is uncontrolled despite adherence with maximal optimized therapy and treatment contributory factors or that worsens when high dose treatment is reduced.
  2. Globally. over 260 million people had poorly controlled asthma highest rate on Australia.3-3-Heart diseases are the most common cause of
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-17 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To Evaluation of cardiac burden in patients with sever bronchial asthma | Baseline
  For Early detection and avoidance of cardiac effects in severe asthma patients